CLINICAL TRIAL: NCT00541619
Title: Sympathetic Overactivity in Essential Hypertension
Status: Withdrawn | Type: Observational
Why Stopped: No patients could be recruited.
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: RE-No.3210
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension; Proteinuria
Keywords: hypertension; sympathetic activity; early renal damage
MeSH Terms: conditions — Hypertension; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- A: hypertensives with proteinuria

SUMMARY:
The primary objective of the study is whether subjects with hypertension and proteinuria display increased sympathetic nerve activity compared to hypertensive subjects without proteinuria and normotensive controls.

ELIGIBILITY:
Inclusion Criteria:

* Normotension or hypertension

Exclusion Criteria:

* Pregnant and nursing women
* Myocardial infarction, clinical signs of coronary heart disease
* Severe depression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary hypertension.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Veelken, MD, Principal Investigator — Principal Investigator
Locations (1):
- Nephrology and Hypertension, Clinical Research Center, Erlangen, Bavaria, Germany